CLINICAL TRIAL: NCT04659876
Title: Clinical Characteristics and Laboratory Values Affecting Mortality in Critical Coronavirus Disease 2019 Patients Followed in the Intensive Care Unit
Brief Title: Factors Affecting Mortality in Critical Patients Admitted to Intensive Care Unit Due to Coronavirus Disease 2019
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Osman Uzundere, Anesthesiology and reanimation specialist, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Other Study IDs: September 11, 2020: 550
Record Dates: First submitted 2020-12-08; First posted 2020-12-09 (Actual); Results first posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Covid19 and Mortality
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Grup S (Survivors): Survivors in ICU follow-up
  Interventions: Diagnostic Test: clinical features and laboratory values
- Grup NS (Nonsurvivors): Patients who died in ICU follow-up
  Interventions: Diagnostic Test: clinical features and laboratory values

INTERVENTIONS:
Diagnostic Test: clinical features and laboratory values — Patients' age, gender, comorbidity, APACHE II, SOFA and KDIGO scores when first admitted to the ICU, performing hemogram (WBC, neutrophil, lymphocyte, neutrophil / lymphocyte ratio, hemoglobin, hematocrit, platelet count), blood gas information (pH, PO2, PCO2, HCO3, lactate), coagulation parameters PTZ and D-dimer, blood biochemistry results (CRP, LDH, CK, urea, creatinine, ALT, AST, total bilirubin, direct bilirubin and indirect bilirubin), procalcitonin and ferritin levels will be recorded. In addition, the number of days spent in the ICU and whether mortality develops or not will be recorded.

SUMMARY:
Gazi Yasargil Training and Research Hospital, located in Diyarbakır province in southeastern Turkey, was designed as a pandemic hospital from the beginning of the coronavirus disease-2019 (COVID-19) outbreak. The first cases in this region were seen on March 22, 2020. In this study, it is aimed to retrospectively examine critical patients admitted to the intensive care unit (ICU) due to COVID-19 from the first onset of cases until September 01, 2020 and to examine the factors affecting mortality. The necessary permits for the study were obtained from the Scientific Research Platform of the T.R. Ministry of Health and the Ethics Committee of the Gazi Yasargil educational and Research Hospital in Diyarbakır. (No: 550, 11.09.2020) Patients diagnosed with COVID-19 on the specified dates, followed in the ICU, older than 18 years, identified as critical/serious according to the World Health Organization and provisional guidelines of the Scientific Board of the T.R. Ministry of Health will be included in the study.

ICU patients without COVID-19; COVID-19 patients under 18 years of age; COVID-19 patients with mild to moderate symptoms, no respiratory distress, no signs of common pneumonia on lung radiography or tomography will be excluded from the study.

Patients' age, gender, comorbidity, Acute Physiology and Chronic Health Evaluation II (APACHE II), Sequential Organ Failure Assessment (SOFA) and Kidney Disease: Improving Global Outcomes (KDIGO) scores when first admitted to the ICU, hemogram parameters (white blood cell count, neutrophil, lymphocyte, neutrophil / lymphocyte ratio, hemoglobin, hematocrit, platelet count), blood gas information (pH, Partial oxygen pressure-PO2, Partial pressure of carbon dioxide-PCO2, bicarbonate-HCO3, lactate), coagulation parameters (prothrombin time and D-dimer, blood biochemistry results (C-reactive protein, lactate dehydrogenase, creatine kinase , urea, creatinine, alanine aminotransferase, aspartate aminotransferase, total bilirubin, direct bilirubin and indirect bilirubin), procalcitonin and ferritin levels will be recorded. In addition, the number of days spent in the ICU and whether mortality develops or not will be recorded.

Patients will be divided into two groups according to their clinical results as those without mortality during ICU follow-up (Group S) and those with mortality (Group NS). The clinical characteristics of both groups, APACHE II, SOFA, KDIGO scores and laboratory results at the first admission to the ICU will be compared. With the diagnosis of COVID-19, factors affecting mortality in critical patients in the ICU will be tried to be determined.

ELIGIBILITY:
Inclusion Criteria:

* During the period between 22.03.2020 and 01.09.2020, critical patients over the age of 18 who were admitted to the ICU of Diyarbakır Gazi Yasargil Educational and Research Hospital due to COVID-19 will be included in the study.

Exclusion Criteria:

* ICU patients without COVID-19
* COVID-19 patients under 18 years of age
* COVID-19 patients with mild to moderate symptoms, no respiratory distress, no signs of common pneumonia on lung radiography or tomography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critical patients over the age of 18 who were admitted to the ICU
Sampling Method: Non-Probability Sample
Enrollment: 445 (Actual)
Dates: Start 2020-03-22 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-12-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Diyarbakır Gazi Yaşargil Training and Research Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mehraeen E, Karimi A, Barzegary A, Vahedi F, Afsahi AM, Dadras O, Moradmand-Badie B, Seyed Alinaghi SA, Jahanfar S. Predictors of mortality in patients with COVID-19-a systematic review. Eur J Integr Med. 2020 Dec;40:101226. doi: 10.1016/j.eujim.2020.101226. Epub 2020 Oct 17. PMID 33101547
- [Background] Luo M, Cao S, Wei L, Zhao X, Gao F, Li S, Meng L, Wang Y. Intubation, mortality, and risk factors in critically ill Covid-19 patients: A pilot study. J Clin Anesth. 2020 Dec;67:110039. doi: 10.1016/j.jclinane.2020.110039. Epub 2020 Sep 7. No abstract available. PMID 32920347
- [Background] Linli Z, Chen Y, Tian G, Guo S, Fei Y. Identifying and quantifying robust risk factors for mortality in critically ill patients with COVID-19 using quantile regression. Am J Emerg Med. 2021 Jul;45:345-351. doi: 10.1016/j.ajem.2020.08.090. Epub 2020 Sep 3. PMID 33046291

RESULTS

PARTICIPANT FLOW:
Groups:
- Grup S (Survivors): Survivors in ICU follow-up
  clinical features and laboratory values: Patients' age, gender, comorbidity, ABO and Rh blood groups, APACHE II, SOFA and KDIGO scores when first admitted to the ICU, performing hemogram (WBC, neutrophil, lymphocyte, neutrophil / lymphocyte ratio, hemoglobin, hematocrit, platelet count), blood gas information (pH, PO2, PCO2, HCO3, lactate), coagulation parameters PTZ and D-dimer, blood biochemistry results (CRP, LDH, CK, urea, creatinine, ALT, AST, total bilirubin, direct bilirubin and indirect bilirubin), procalcitonin and ferritin levels will be recorded. In addition, the number of days spent in the ICU and whether mortality develops or not will be recorded.
- Grup NS (Nonsurvivors): Patients who died in ICU follow-up
  clinical features and laboratory values: Patients' age, gender, comorbidity, ABO and Rh blood groups, APACHE II, SOFA and KDIGO scores when first admitted to the ICU, performing hemogram (WBC, neutrophil, lymphocyte, neutrophil / lymphocyte ratio, hemoglobin, hematocrit, platelet count), blood gas information (pH, PO2, PCO2, HCO3, lactate), coagulation parameters PTZ and D-dimer, blood biochemistry results (CRP, LDH, CK, urea, creatinine, ALT, AST, total bilirubin, direct bilirubin and indirect bilirubin), procalcitonin and ferritin levels will be recorded. In addition, the number of days spent in the ICU and whether mortality develops or not will be recorded.
Period: Overall Study
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Started | 149 | 296
Completed | 149 | 296
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors) | Total
Number analyzed (Participants) | 149 | 296 | 445
Age, Continuous [Mean (Full Range); unit: years] | 62.7 [22 to 95] | 71.4 [18 to 100] | 68.5 [18 to 100]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 130 | 213
  Male | 66 | 166 | 232
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Comorbidity [Count of Participants; unit: Participants]
  No | 42 | 65 | 107
  Yes | 107 | 231 | 338

OUTCOME MEASURES:

1. Primary Outcome: Acute Physiology and Chronic Health Evaluation II Score
Description: The score can help in the assessment of patients to determine the level & degree of diagnostic & therapeutic intervention.
  Interpretation of APACHE II: minimum 0 and maximum 71; increasing score is associated with an increasing risk of hospital death.
Time Frame: APACHE II score on the first admission of ICU
Population: APACHE II score
Measure: Mean (Full Range); unit: score on a scale
Groups:
- APACHE II Score Grup S (Survivors): Survivors in ICU follow-up
  clinical features and laboratory values: Patients' age, gender, comorbidity, ABO and Rh blood groups, APACHE II, SOFA and KDIGO scores when first admitted to the ICU, performing hemogram (WBC, neutrophil, lymphocyte, neutrophil / lymphocyte ratio, hemoglobin, hematocrit, platelet count), blood gas information (pH, PO2, PCO2, HCO3, lactate), coagulation parameters PTZ and D-dimer, blood biochemistry results (CRP, LDH, CK, urea, creatinine, ALT, AST, total bilirubin, direct bilirubin and indirect bilirubin), procalcitonin and ferritin levels will be recorded. In addition, the number of days spent in the ICU and whether mortality develops or not will be recorded.
- APACHE II Score Grup NS (Nonsurvivors): Patients who died in ICU follow-up
  clinical features and laboratory values: Patients' age, gender, comorbidity, ABO and Rh blood groups, APACHE II, SOFA and KDIGO scores when first admitted to the ICU, performing hemogram (WBC, neutrophil, lymphocyte, neutrophil / lymphocyte ratio, hemoglobin, hematocrit, platelet count), blood gas information (pH, PO2, PCO2, HCO3, lactate), coagulation parameters PTZ and D-dimer, blood biochemistry results (CRP, LDH, CK, urea, creatinine, ALT, AST, total bilirubin, direct bilirubin and indirect bilirubin), procalcitonin and ferritin levels will be recorded. In addition, the number of days spent in the ICU and whether mortality develops or not will be recorded.
Arm/Group | APACHE II Score Grup S (Survivors) | APACHE II Score Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
score on a scale | 13.1 [2 to 33] | 18.3 [2 to 49]

2. Primary Outcome: Sequential Organ Failure Assessment Score
Description: The Sequential Organ Failure Assessment (SOFA) score is a scoring system that assesses the performance of several organ systems in the body (neurologic, blood, liver, kidney, and blood pressure/hemodynamics) and assigns a score based on the data obtained in each category. The SOFA score is made of 6 variables, each representing an organ system. Each organ system is assigned a point value from 0 (normal) to 4 (high degree of dysfunction/failure). Score ranges from 0 (best) to 24 (worst) points.
Time Frame: SOFA score on the first admission of ICU
Measure: Mean (Full Range); unit: units on a scale
Groups:
- SOFA Score Grup S (Survivors): Survivors in ICU follow-up
  clinical features and laboratory values: Patients' age, gender, comorbidity, ABO and Rh blood groups, APACHE II, SOFA and KDIGO scores when first admitted to the ICU, performing hemogram (WBC, neutrophil, lymphocyte, neutrophil / lymphocyte ratio, hemoglobin, hematocrit, platelet count), blood gas information (pH, PO2, PCO2, HCO3, lactate), coagulation parameters PTZ and D-dimer, blood biochemistry results (CRP, LDH, CK, urea, creatinine, ALT, AST, total bilirubin, direct bilirubin and indirect bilirubin), procalcitonin and ferritin levels will be recorded. In addition, the number of days spent in the ICU and whether mortality develops or not will be recorded.
- SOFA Score Grup NS (Nonsurvivors): Patients who died in ICU follow-up
  clinical features and laboratory values: Patients' age, gender, comorbidity, ABO and Rh blood groups, APACHE II, SOFA and KDIGO scores when first admitted to the ICU, performing hemogram (WBC, neutrophil, lymphocyte, neutrophil / lymphocyte ratio, hemoglobin, hematocrit, platelet count), blood gas information (pH, PO2, PCO2, HCO3, lactate), coagulation parameters PTZ and D-dimer, blood biochemistry results (CRP, LDH, CK, urea, creatinine, ALT, AST, total bilirubin, direct bilirubin and indirect bilirubin), procalcitonin and ferritin levels will be recorded. In addition, the number of days spent in the ICU and whether mortality develops or not will be recorded.
Arm/Group | SOFA Score Grup S (Survivors) | SOFA Score Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
units on a scale | 3.3 [1 to 12] | 4.8 [1 to 17]

3. Primary Outcome: Kidney Disease: Improving Global Outcomes Scores
Description: It is a system used to determine the severity of kidney failure. It is a classification consisting of four stages: 0-1-2-3. It indicates that the level of failure worsens as the stage increases.
Time Frame: When the patients were admitted to ICU for the first time.
Measure: Count of Participants; unit: Participants
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
Participants
  KDIGO 0 | 113 | 76
  KDIGO 1 | 17 | 66
  KDIGO 2 | 12 | 67
  KDIGO 3 | 7 | 87

4. Primary Outcome: White Blood Cell
Description: White blood cell count was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: At ICU admission
Population: All participants included in the study were analyzed for this outcome. The numbers analyzed are identical to those reported in the participant flow.
Measure: Mean (Full Range); unit: cells × 10³/µL
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
cells × 10³/µL | 10.6 [2.95 to 42.7] | 11.6 [1.13 to 57.4]

5. Primary Outcome: Neutrophil
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: When the patients were admitted to ICU for the first time
Population: as for outcome 4
Measure: Mean (Full Range); unit: cells × 10³/µL
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
cells × 10³/µL | 8.75 [1.3 to 37.5] | 9.9 [0.66 to 34.4]

6. Primary Outcome: Lymphocyte
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: When the patients were admitted to ICU for the first time
Population: as for outcome 4
Measure: Mean (Full Range); unit: cells × 10³/µL
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
cells × 10³/µL | 1.1 [0.19 to 3.59] | 0.93 [0.14 to 3.5]

7. Primary Outcome: Neutrophil Lymphocyte Ratio
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: the first admission to ICU
Population: as for outcome 4
Measure: Mean (Full Range); unit: Ratio
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
Ratio | 9.4 [0.33 to 60.04] | 14.5 [0.12 to 87.1]

8. Primary Outcome: Comorbidities
Description: The presence of this comorbidity was determined based on medical history documented in medical records at ICU admission.
Time Frame: When the patients were admitted to ICU for the first time
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
Participants
  No | 42 | 65
  Yes | 107 | 231

9. Primary Outcome: Diabetes
Description: The presence of this comorbidity was determined based on medical history documented in medical records at ICU admission.
Time Frame: When the patients were admitted to ICU for the first time
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
Participants | 38 | 89

10. Primary Outcome: Hypertension
Description: The presence of this comorbidity was determined based on medical history documented in medical records at ICU admission.
Time Frame: When the patients were admitted to ICU for the first time
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
Participants | 64 | 114

11. Primary Outcome: Chronic Obstructive Pulmonary Disease
Description: The presence of this comorbidity was determined based on medical history documented in medical records at ICU admission.
Time Frame: When the patients were admitted to ICU for the first time
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
Participants | 19 | 26

12. Primary Outcome: Chronic Kidney Disease
Description: The presence of this comorbidity was determined based on medical history documented in medical records at ICU admission.
Time Frame: When the patients were admitted to ICU for the first time
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
Participants | 12 | 22

13. Primary Outcome: Cardiovascular Disease
Description: The presence of this comorbidity was determined based on medical history documented in medical records at ICU admission.
Time Frame: When the patients were admitted to ICU for the first time
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
Participants | 19 | 47

14. Primary Outcome: Hemoglobin
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: At ICU admission (first laboratory measurement after ICU admission)
Population: as for outcome 4
Measure: Mean (Full Range); unit: g/dl
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
g/dl | 13.06 [5.9 to 17] | 12.6 [5.6 to 19.2]

15. Primary Outcome: Hematocrit
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: At ICU admission (first laboratory measurement after ICU admission)
Population: as for outcome 4
Measure: Mean (Full Range); unit: percentage of red blood cell
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
percentage of red blood cell | 40.61 [17.8 to 61.6] | 41.2 [20.2 to 55.9]

16. Primary Outcome: Platelet
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: At ICU admission (first laboratory measurement after ICU admission)
Population: as for outcome 4
Measure: Mean (Full Range); unit: ×1000/uL
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
×1000/uL | 253.4 [84 to 671] | 237.3 [30 to 628]

17. Primary Outcome: Prothrombin Time
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: At ICU admission (first laboratory measurement after ICU admission)
Population: as for outcome 4
Measure: Mean (Full Range); unit: second
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
second | 13.3 [9.9 to 22.5] | 14.1 [9.7 to 54.9]

18. Primary Outcome: D-dimer
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: At ICU admission (first laboratory measurement after ICU admission)
Population: as for outcome 4
Measure: Mean (Full Range); unit: ng/ml
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
ng/ml | 954.5 [75 to 16948] | 2564.4 [8.4 to 44498]

19. Primary Outcome: Blood Gas Analysis-pH
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: At ICU admission (first laboratory measurement after ICU admission)
Population: as for outcome 4
Measure: Mean (Full Range); unit: Quantitative measure of the acidity
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
Quantitative measure of the acidity | 7.38 [6.91 to 7.54] | 7.36 [6.82 to 7.55]

20. Primary Outcome: Partial Oxygen Pressure
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: At ICU admission (first laboratory measurement after ICU admission)
Population: as for outcome 4
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
mmHg | 42.14 [17.9 to 162] | 40.3 [13.5 to 198]

21. Primary Outcome: Partial Pressure of Carbon Dioxide
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: At ICU admission (first laboratory measurement after ICU admission)
Population: as for outcome 4
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
mmHg | 39.1 [16.9 to 108] | 38.61 [20 to 115]

22. Primary Outcome: Bicarbonate
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: At ICU admission (first laboratory measurement after ICU admission)
Population: as for outcome 4
Measure: Mean (Full Range); unit: mmol/L
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
mmol/L | 23.02 [5.9 to 31.5] | 21.16 [5.3 to 32.1]

23. Primary Outcome: Lactate
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: At ICU admission (first laboratory measurement after ICU admission)
Population: as for outcome 4
Measure: Mean (Full Range); unit: mmol/L
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
mmol/L | 2.2 [0.6 to 8.2] | 3.04 [0.7 to 26]

24. Primary Outcome: Lactate Dehydrogenase
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: At ICU admission (first laboratory measurement after ICU admission)
Population: as for outcome 4
Measure: Mean (Full Range); unit: U/L
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
U/L | 406.7 [139 to 1079] | 569.4 [99 to 4500]

25. Primary Outcome: Creatine Kinase
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: At ICU admission (first laboratory measurement after ICU admission)
Population: as for outcome 4
Measure: Mean (Full Range); unit: IU/L
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
IU/L | 204.4 [11 to 2949] | 369.4 [0.32 to 14952]

26. Primary Outcome: C-reactive Protein
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: At ICU admission (first laboratory measurement after ICU admission)
Population: as for outcome 4
Measure: Mean (Full Range); unit: mg/L
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
mg/L | 120.4 [2 to 350] | 151.7 [2 to 350]

27. Primary Outcome: Blood Urea Nitrogen
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: At ICU admission (first laboratory measurement after ICU admission)
Population: as for outcome 4
Measure: Mean (Full Range); unit: mg/dl
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
mg/dl | 47.6 [8 to 267] | 72.5 [13 to 280]

28. Primary Outcome: Creatinine
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: At ICU admission (first laboratory measurement after ICU admission)
Population: as for outcome 4
Measure: Mean (Full Range); unit: mg/dl
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
mg/dl | 1.28 [0.44 to 10.4] | 1.68 [0.36 to 21.8]

29. Primary Outcome: Alanine Aminotransferase
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: At ICU admission (first laboratory measurement after ICU admission)
Population: as for outcome 4
Measure: Mean (Full Range); unit: U/L
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
U/L | 32.2 [6 to 442] | 47.9 [6 to 1254]

30. Primary Outcome: Aspartate Aminotransferase
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: At ICU admission (first laboratory measurement after ICU admission)
Population: as for outcome 4
Measure: Mean (Full Range); unit: U/L
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
U/L | 40.8 [9 to 518] | 81.5 [7 to 3444]

31. Primary Outcome: Total Bilirubin
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: At ICU admission (first laboratory measurement after ICU admission)
Population: as for outcome 4
Measure: Mean (Full Range); unit: mg/dl
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
mg/dl | 0.68 [0.14 to 3.69] | 0.75 [0.12 to 6.8]

32. Primary Outcome: Direct Bilirubin
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: At ICU admission (first laboratory measurement after ICU admission)
Population: as for outcome 4
Measure: Mean (Full Range); unit: mg/dl
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
mg/dl | 0.34 [0.1 to 2.31] | 0.4 [0.1 to 4.7]

33. Primary Outcome: Indirect Bilirubin
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: At ICU admission (first laboratory measurement after ICU admission)
Population: as for outcome 4
Measure: Mean (Full Range); unit: mg/dl
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
mg/dl | 0.33 [0.03 to 1.86] | 0.33 [0.01 to 2]

34. Primary Outcome: Procalcitonin
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: At ICU admission (first laboratory measurement after ICU admission)
Population: as for outcome 4
Measure: Mean (Full Range); unit: ng/ml
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
ng/ml | 1.39 [0.02 to 62.8] | 4.13 [0.03 to 100]

35. Primary Outcome: Ferritin
Description: This parameter was measured using routinely collected laboratory data obtained from medical records at ICU admission.
Time Frame: At ICU admission (first laboratory measurement after ICU admission)
Population: as for outcome 4
Measure: Mean (Full Range); unit: μg/L
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
μg/L | 673.8 [5.86 to 2000] | 951.5 [16.6 to 2000]

36. Secondary Outcome: Length of Stay in the Intensive Care Unit
Description: ICU length of stay was measured as the total number of days from ICU admission to ICU discharge or death, based on information recorded in medical records.
Time Frame: Three months
Population: as for outcome 4
Measure: Mean (Full Range); unit: Day
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
Number analyzed (Participants) | 149 | 296
Day | 13.02 [1 to 91] | 10.3 [1 to 79]

ADVERSE EVENTS:
Time Frame: During ICU stay
Description: This was a retrospective observational study. All-cause mortality was systematically assessed using medical records during the ICU stay. Other adverse events were not systematically collected or analyzed.
Arm/Group | Grup S (Survivors) | Grup NS (Nonsurvivors)
All-Cause Mortality (participants affected / at risk) | 0/149 | 296/296
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT04659876/Prot_SAP_000.pdf